CLINICAL TRIAL: NCT06590935
Title: Prospective Cohort Study on Endocrine and Exocrine Secretory Function Alterations After Moderately Severe and Severe Acute Pancreatitis
Brief Title: Endocrine and Exocrine Secretory Function Alterations After Moderately Severe and Severe Acute Pancreatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Other Study IDs: NMU-3cDM-1B
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Acute Pancreatitis (AP); Diabetes Mellitus
Keywords: Acute pancreatitis; Diabetes mellitus; PPDM-A; Risk factor
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected at every visit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute pancreatitis: Patients with a complete diagnosis of MSAP and SAP

SUMMARY:
The goal of this observational study is to learn about post-acute pancreatitis diabetes mellitus (PPDM-A). The main questions it aims to answer are:

1. Are the incident rates of glucose metabolic disorders (pre-diabetes and diabetes mellitus) after acute pancreatitis of different etiologies the same?
2. Are alterations in endocrine and exocrine secretory function in patients with acute pancreatitis associated with all-round outcomes?

All patients with acute pancreatitis have been given the standardized treatment for the condition.

Investigators will compare the incident rates of glucose metabolic disorders (pre-diabetes and diabetes mellitus) after acute pancreatitis of different etiologies in patients with moderately severe (MSAP) and severe acute pancreatitis (SAP) to explore the association between alterations in endocrine and exocrine secretory function and all-round outcomes.

DETAILED DESCRIPTION:
Investigators will prospectively collect data from patients with moderately severe (MSAP) and severe acute pancreatitis (SAP) in participant centers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Chinese subjects;
2. Age ≥18 years at the time of signing the informed consent;
3. Patients with a complete diagnosis of MSAP and SAP (according to the Chinese guidelines for the diagnosis and treatment of acute pancreatitis 2019);
4. Voluntary signatories of informed consent

Exclusion Criteria:

1. Patients with a history of diabetes mellitus or pre-diabetes mellitus, or glycosylated hemoglobin ≥ 6.0% or venous FPG ≥ 6.1 mmol/L at admission;
2. Patients have any evidence of type 1 diabetes-related autoimmunity;
3. Patients have any risk for secondary diabetes due to exposure to medications or other endocrine diseases;
4. Combined with pancreas-related trauma or a history of pancreatic surgery;
5. Patients undergo pancreatic surgery during treatment;
6. Pregnancy or breastfeeding;
7. Patients suffer from severe cardiac, hepatic or renal insufficiency or malignant diseases;
8. Failure to sign informed consent due to cognitive impairment or other conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will collect data from patients with moderately severe (MSAP) and severe acute pancreatitis (SAP) in participant centers.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who developed glucose metabolic disorders (pre-diabetes and diabetes mellitus) | From the AP treatment to 5 years after the end of treatment
  The diagnosis of glucose metabolic disorders should be made applying the criteria of the American Diabetes Association.

CONTACTS AND LOCATIONS:
Overall Officials: Tuo Li, Prof., Study Director — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bharmal SH, Cho J, Ko J, Petrov MS. Glucose variability during the early course of acute pancreatitis predicts two-year probability of new-onset diabetes: A prospective longitudinal cohort study. United European Gastroenterol J. 2022 Mar;10(2):179-189. doi: 10.1002/ueg2.12190. Epub 2022 Feb 20. PMID 35188346
- [Background] Bharmal SH, Cho J, Alarcon Ramos GC, Ko J, Stuart CE, Modesto AE, Singh RG, Petrov MS. Trajectories of glycaemia following acute pancreatitis: a prospective longitudinal cohort study with 24 months follow-up. J Gastroenterol. 2020 Aug;55(8):775-788. doi: 10.1007/s00535-020-01682-y. Epub 2020 Jun 3. PMID 32494905
- [Background] Zhong S, Du Q, Liu N, Chen Y, Yang T, Qin S, Jiang Y, Huang X. Developing a CT-based radiomics nomogram for predicting post-acute pancreatitis diabetes mellitus incidence. Br J Radiol. 2023 Dec;96(1152):20230382. doi: 10.1259/bjr.20230382. Epub 2023 Oct 24. PMID 37750855
- [Background] Lv Y, Zhang J, Yang T, Sun J, Hou J, Chen Z, Yu X, Yuan X, Lu X, Xie T, Yu T, Su X, Liu G, Zhang C, Li L. Non-Alcoholic Fatty Liver Disease (NAFLD) Is an Independent Risk Factor for Developing New-Onset Diabetes After Acute Pancreatitis: A Multicenter Retrospective Cohort Study in Chinese Population. Front Endocrinol (Lausanne). 2022 May 25;13:903731. doi: 10.3389/fendo.2022.903731. eCollection 2022. PMID 35692404
- [Background] Yu BJ, Li NS, He WH, He C, Wan JH, Zhu Y, Lu NH. Pancreatic necrosis and severity are independent risk factors for pancreatic endocrine insufficiency after acute pancreatitis: A long-term follow-up study. World J Gastroenterol. 2020 Jun 21;26(23):3260-3270. doi: 10.3748/wjg.v26.i23.3260. PMID 32684740
- [Background] Zhi M, Zhu X, Lugea A, Waldron RT, Pandol SJ, Li L. Incidence of New Onset Diabetes Mellitus Secondary to Acute Pancreatitis: A Systematic Review and Meta-Analysis. Front Physiol. 2019 May 31;10:637. doi: 10.3389/fphys.2019.00637. eCollection 2019. PMID 31231233
- [Background] Das SL, Singh PP, Phillips AR, Murphy R, Windsor JA, Petrov MS. Newly diagnosed diabetes mellitus after acute pancreatitis: a systematic review and meta-analysis. Gut. 2014 May;63(5):818-31. doi: 10.1136/gutjnl-2013-305062. Epub 2013 Aug 8. PMID 23929695
- [Background] Shen HN, Yang CC, Chang YH, Lu CL, Li CY. Risk of Diabetes Mellitus after First-Attack Acute Pancreatitis: A National Population-Based Study. Am J Gastroenterol. 2015 Dec;110(12):1698-706. doi: 10.1038/ajg.2015.356. Epub 2015 Nov 3. PMID 26526084